CLINICAL TRIAL: NCT06418893
Title: Effect of Isoflurane and Target Control Infusion (TCI) Propofol on Intra-operative Usage of Vasopressors in Liver Transplant Recipients: A Randomized Controlled Trial.
Brief Title: Effect of TCI Propofol on Liver Transplant (TCI) Propofol on Intra-operative Usage of Vasopressors in Liver Transplant Recipients.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Collaborators: Institute of Liver and Biliary Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IEC/2023/100/MA05
Record Dates: First submitted 2024-04-17; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Liver Transplant Recipients

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, double blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isoflurane (Active Comparator): Drug- Isoflurane Dosage form- Inhalational, 1-2% Frequency- Continuously Duration- Throughout Intraoperative period
  Interventions: Drug: Inhalational isoflurane
- Propofol (Experimental): Drug- Propofol Dosage form- Intravenously, 2.5 mcg/ml target plasma concentration Frequency- Continuously Duration- Throughout Intraoperative period
  Interventions: Drug: Target control infusion propofol

INTERVENTIONS:
Drug: Target control infusion propofol — target control infusion of propofol for target plasma concentration 2.5mcg/ml and BIS 40-60
  Arms: Propofol
Drug: Inhalational isoflurane — Inhalational Isoflurane at concentration 1-2%
  Arms: Isoflurane

SUMMARY:
Both isoflurane and propofol are being used to give anaesthesia for living donor liver transplant in our institute. Propofol when compared to isoflurane has advantages like early awakening from anaesthesia, reduced nausea, vomiting in the postoperative period. Propofol also has antioxidant properties. Because of its antioxidant properties propofol may have a protective effect against oxidative stress and ischemia reperfusion injury in major organs during liver transplant surgery. However, there are no studies showing the effect of isoflurane and propofol on Intraoperative hemodynamics and postoperative liver and kidney functions.Thus, we are conducting this study to know the effect of these agents on intraoperative hemodynamics and postoperative liver and kidney function.

ELIGIBILITY:
Inclusion Criteria:-Above 18 years of age who will undergo living donor liver transplant

-

Exclusion Criteria: Refusal to consent

* Acute liver failure, Acute on chronic liver failure
* Allergic to propofol or any component of propofol
* Patients with pre existing cardiac dysfunction and cardiomyopathy
* Patients with pre existing renal dysfunction/ deranged RFTs preoperatively

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of total Noradrenaline and vasopressin requirement between isoflurane and TCI propofol group in Living donor liver transplant recipients intraoperatively. | INTRAOPERATIVELY
  TCI propofol will provide more stable hemodynamics

SECONDARY OUTCOMES:
To compare between the two groups mean arterial pressure during different phases of liver transplant recorded every 15 minutes | INTRAOPERATIVELY AT 15 MINUTES INTERVAL
To compare between the two groups mean systemic vascular resistance during different phases of liver transplant recorded every 15 minutes | INTRAOPERATIVELY AT 15 MINUTES INTERVAL
To compare between the two groups cardiac output during different phases of liver transplant recorded every 15 minutes | INTRAOPERATIVELY AT 15 MINUTES INTERVAL
Total vasopressor requirement during reperfusion | Intraoperative
Peak dose of nordrenaline and vasopressin during different phases of liver transplant intraoperatively | Intraoperatively
QTc interval between the two groups during different phases of liver transplant measured every 15 minutes | Intraoperatively every 15 mins
Peak lactate levels intraoperatively | Intraoperatively
Postoperative Liver function tests ie Bilirubin and albumin | at 12, 24, 72 hours and day 7 postoperatively
Postoperative Liver function tests ie AST and ALT | at 12, 24, 72 hours and day 7 postoperatively
Postoperative Liver function tests ie GGT | at 12, 24, 72 hours and day 7 postoperatively
Postoperative Liver function tests ie platelet count | at 12, 24, 72 hours and day 7 postoperatively
Postoperative coagulation profile | at 12, 24, 72 hours and day 7 postoperatively
Postoperative Renal function tests i.e. Blood urea and S.creatinine levels | at12, 24, 72 hours and day7 postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and biliary sciences, Delhi, India

IPD SHARING:
Plan to Share IPD: No